CLINICAL TRIAL: NCT02249299
Title: The Effects of Sativex on Neurocognitive and Behavioural Function in Adults With Attention-deficit/Hyperactivity Disorder; The EMA-C Study (Experimental Medicine in ADHD - Cannabinoids)
Brief Title: Experimental Medicine in ADHD - Cannabinoids
Acronym: EMA-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EMA-C
Record Dates: First submitted 2014-09-03; First posted 2014-09-25 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2015-09

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD,; Cannabis,; Sativex,; Endocannabinoid,; Cognition
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex Oromucosal Spray (Active Comparator): Participants will titrate onto Sativex during the first two weeks of the study, carried out according to a standardised dosing schedule. After 2 weeks the clinician and participant will decide on the optimal dose for the remainder of the 4 week trial
  Interventions: Drug: Sativex Oromucosal Spray
- Placebo (Placebo Comparator): Participants will titrate onto the placebo during the first two weeks of the study, carried out according to a standardised dosing schedule. After 2 weeks the clinician and participant will decide on the optimal dose for the remainder of the 4 week trial
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex Oromucosal Spray — Sativex Oromucosal Spray (GW Pharma Ltd, Salisbury. UK). Each 100 microlitre spray contains: 2.7 mg delta-9-tetrahydrocannabinol (THC) and 2.5 mg cannabidiol (CBD).
  Other Names: Sativex
  Arms: Sativex Oromucosal Spray
Drug: Placebo
  Arms: Placebo

SUMMARY:
Adult patients with ADHD commonly report an improvement in behavioural symptoms when using cannabis with some reporting a preference towards cannabis over their ADHD stimulant medication. The EMA-C study aims to investigate the effects of a cannabis based medication, Sativex Oromucosal Spray on behaviour and cognition in adults with ADHD.

This will be carried out by conducting a placebo controlled trial. 30 adults with ADHD will take Sativex or a dummy medication (a placebo) every day for 6 weeks. There is a 50% chance of receiving the Sativex or Placebo. Measures of behaviour and cognition will be taken before and after 6 weeks of treatment. We hypothesise that treatment with Sativex will result in improvements in behaviour and cognition above that of the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* The study is open for both men and women aged 18-55 who meet DSM 5 criteria for ADHD (N= 30). Subjects will be either unmedicated or medicated with stimulant medication only and be willing to come of this medication for 1 week before and for the duration of the study. To ensure that this does not disadvantage patients we will only include those on stimulant medication who do not take medication on a regular basis and where short periods of medication are not thought by both the patient and psychiatrist to represent a clinical problem in the overall control of the symptoms and impairments. For example, by including patients who are considering a "stimulant drug holiday", which is a common clinical procedure in ADHD. Subjects must not use other prescription and non-prescription medication or recreational drugs during the study.

Exclusion Criteria:

* Exclusion criteria will include autism spectrum disorders and other psychiatric disorders including recurrent major depression, bipolar I disorder, any psychotic disorder and obsessive compulsive disorder and learning difficulties defined as an IQ < 70. Neurological problems and known or suspected history of a drug or alcohol dependence disorder. Subjects who are using or have used cannabis or cannabis based medications in the 30 day period prior to study entry. Concurrent history of renal, hepatic, cardiovascular or convulsive disorders. Females who are pregnant or breastfeeding. Female subjects of child bearing potential and male subjects whose partner is of child bearing potential, unless willing to ensure that they or their partner use two effective forms of contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for three months thereafter (Note: a male condom should not be used in conjunction with a female condom).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in performance on the QB Test using the average of 3 weighted indexes: 'activity' 'inattention' and 'impulsivity' | 6 weeks (baseline (day 1)-follow-up (day 42))
  QbTest: The Qb test is a computer administered attention test. An infrared camera monitors patient movement and measures activity; attention and impulsivity are calculated based on the task performance and activity level. The data is processed and compared with a normative group.

SECONDARY OUTCOMES:
ADHD symptoms of inattention, hyperactivity-impulsivity and emotional lability | 6 weeks (baseline (day 1) - follow-up (day 42))
  This will be assessed using the Conners' Adult ADHD Rating Scales (CAARS) and Wender-Reimher Adult Attention Deficit Disorder Scale (WRAADS) combined (investigator rated): Both measure ADHD symptom severity.
Self-report behavioural questionnaire | 6 weeks (baseline (day 1) - follow-up (day 42)
  Executive function measured with: The Brief-A.
Self-report behavioural questionnaire | 6 weeks (baseline (day 1) - follow-up (day 42)
  Common psychopathology measured with: The Symptom Check-List (SCL-90)
Self-report behavioural questionnaire | 6 weeks (baseline (day 1) - follow-up (day 42)
  Mood will be measured using: The Centre for Neurologic Studies-Lability Scale (CNS-LS)
Self-report behavioural questionnaire | 6 weeks (baseline (day 1) - follow-up (day 42)
  Mood measured with: The Affective Lability Scale (ALS-SF)
Self-report behavioural questionnaires | 6 weeks (baseline (day 1) - follow-up (day 42)
  Sleep measured with: The Pittsburgh Sleep Quality Index (PSQI)
Self-report behavioural questionnaire | 6 weeks (baseline (day 1) - follow-up (day 42)
  Level of depressive thoughts: The Depressive Thoughts Questionnaire (DTQ)
Self-report behavioural questionnaire | 6 weeks (baseline (day 1) - follow-up (day 42)
  Control over thoughts: Cognitive Control Questionnaire
Self-report behavioural questionnaire | 6 weeks (baseline (day 1) - follow-up (day 42)
  The Brief COPE assesses how participants are coping with stressful life events
Self-report behavioural questionnaire | 6 weeks (baseline (day 1) - follow-up (day 42)
  The Brief Life Events Questionnaire (BLEQ) assesses the occurrence of stressful life events.
Self-report behavioural questionnaires | 6 weeks (baseline (day 1) - follow-up (day 42)
  Functional Impairment: The Weiss Functional Impairment Rating Scale Self Report (WFIRS-S)
Self-report behavioural questionnaires | 6 weeks (baseline (day 1) - follow-up (day 42)
  The Adult ADHD Quality of Life Scales (AAQoL)
Change in cognitive performance | 6 weeks (baseline (day 1)-follow-up (day 42))
  SART: The SART is a computerised go/no go task measuring both response inhibition and sustained attention

CONTACTS AND LOCATIONS:
Overall Officials: Philip Asherson, MD, PhD, Principal Investigator — Institute of Psychiatry, King's College London
Locations (1):
- Social, Genetic and Developmental Psychiatry Centre, Institute of Psychiatry, King's College London, London, United Kingdom

REFERENCES:
- [Result] Cooper RE, Williams E, Seegobin S, Tye C, Kuntsi J, Asherson P. Cannabinoids in attention-deficit/hyperactivity disorder: A randomised-controlled trial. Eur Neuropsychopharmacol. 2017 Aug;27(8):795-808. doi: 10.1016/j.euroneuro.2017.05.005. Epub 2017 May 30. PMID 28576350